CLINICAL TRIAL: NCT04995497
Title: IV vs. Erector Spinae Plane Blocks-Cardiac Surgery
Brief Title: Intravenous(IV) vs. Erector Spinae Plane Blocks in Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Archit Sharma (Other)
Responsible Party: Sponsor-Investigator, Archit Sharma, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202009510
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Erector Spinae Plane Block; Pain Control; Post-Operative Pain, Chronic
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erector Spinae Plane Block-Administration of Lidocaine (Experimental): Bilateral ultrasound guided erector spinae plane catheter placement for the administration of lidocaine. Dose will be 2 mg/kg ideal body weight. Bolus will be divided equally between the two ESP catheters. This is followed by lidocaine infusion via ESP catheter at 2 mg/kg/hr for 48 hours after catheter placement.
  Interventions: Drug: Administration of Lidocaine Post Cardiac Surgery via ESP Catheter
- Intravenous-Administration of Lidocaine (Active Comparator): Subject will receive a bolus of lidocaine at 2 mg/kg ideal body weight. This is followed by lidocaine infusion via intravenous route at 2 mg/kg/hr for 48 hours.
  Interventions: Drug: Intravenous Administration of Lidocaine Post Cardiac Surgery

INTERVENTIONS:
Drug: Intravenous Administration of Lidocaine Post Cardiac Surgery — Lidocaine will be administered via intravenously. Initial dose will be at 2 mg/kg ideal body weight followed by dosing at 2 mg/kg/hr for 48 hours
  Other Names: Pain control post cardiac surgery
  Arms: Intravenous-Administration of Lidocaine
Drug: Administration of Lidocaine Post Cardiac Surgery via ESP Catheter — Lidocaine will be administered via ESP catheter. Initial dose will be at 2 mg/kg ideal body weight split between two catheters followed by dosing at 2 mg/kg/hr for 48 hours
  Other Names: Pain control post cardiac surgery
  Arms: Erector Spinae Plane Block-Administration of Lidocaine

SUMMARY:
Interfascial plane blocks have been developed for analgesia, among which the erector spinae plane (ESP) has gained popularity. The ESP block has been hypothesized to provide truncal analgesia by spread of local anesthetic into the paravertebral space. Recent studies have contested this idea showing unreliability in the spread of the local anesthetic into the paravertebral space.

DETAILED DESCRIPTION:
Post-operative pain is a significant issue following open heart surgeries and poorly controlled pain can result in significant cardiorespiratory morbidity. Many patients suffer pain both at rest (49%) and on movement (62%) following open heart surgeries via sternotomy and adequate pain management requires closer re-assessment and treatment. The intensity of pain is noted to be higher in the first 48 hours post surgery and hence modalities to control pain may make the greatest difference in the first 2 days after surgery.

Enhanced recovery pathways utilizing multimodal analgesia have shown significant analgesic and opioid sparing benefit while minimizing ICU and length of hospital stays. Some multimodal regimens have also incorporated regional blocks but the optimal analgesic regimen remains elusive. The ESP block has been hypothesized to provide truncal anesthesia by spread of local anesthetic into the paravertebral space, but recent studies contest this idea. Bilateral paravertebral blocks can result in higher than acceptable levels of local anesthetic in both cardiac and non-cardiac surgical patients and this may be true following bilateral erector spinae plane (ESP) as well. Hence, the pharmacokinetic profile of administered local anesthetics is necessary given the lack of information about the local anesthetic systemic levels following bilateral ESP.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective cardiac surgery for coronary artery bypass graft (CABG) or valve surgery via sternotomy.
* English speaking

Exclusion Criteria:

* Emergency surgery
* Allergy to medications (ie lidocaine)
* BMI less than 20 or greater than 50
* Major liver or kidney dysfunction or other pre-existing major organ dysfunction
* Revision cardiac surgery
* Surgery via thoracotomy
* Off-pump coronary artery bypass
* Narcotic dependent (Opioid intake morphine equivalents greater than 10mg/day for more than 3 months
* Chronic pain (ie fibromyalgia)
* Significant central nervous system or respiratory disease
* Hematological disorders or de-ranged coagulation parameters
* Psychiatric illness that impedes subject from providing informed consent
* Pre-operative neurological deficits
* Language barrier
* Inability to provide informed consent
* Prisoner status
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2023-04-07 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Archit Sharma, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous-Administration of Lidocaine: Sham block procedure (catheter will be taped to subjects skin). Subject will receive a bolus of lidocaine at 2 mg/kg ideal body weight. This is followed by lidocaine infusion via intravenous route at 2 mg/kg/hr for 48 hours after sham catheter placement.
  Intravenous Administration of Lidocaine Post Cardiac Surgery: Lidocaine will be administered via intravenously. Initial dose will be at 2 mg/kg ideal body weight followed by dosing at 2 mg/kg/hr for 48 hours
Period: Overall Study
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Started | 36 | 34
Completed | 29 | 28
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Population: It is the same.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.36 (10.1) | 67.94 (8.28) | 66.61 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 30 | 28 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 34 | 33 | 67
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 35 | 32 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Quantitate the Amount of Opioid Medication Required to Provide Pain Relief-Cumulative First 48 Hours
Description: To assess if either route (IV or ESP catheter) of lidocaine provided maximal pain relief when compared to its counterpart, the type and amount of medication provided the subject will be recorded. Cumulative opioid usage amounts required to provide relief during the first 48 hours will be tabulated in morphine equivalents. A comparison will be made between the two route to see if one route is optimal over the other. The variables will be presented as median and interquartile range.
Time Frame: 48 hours post surgical intervention
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 30 | 30
Morphine Milligram Equivalents | 80.2 [39.45 to 122.98] | 54.9 [30.88 to 100.83]

2. Primary Outcome: Compare Pain Score Reported by Subject 48 Hours Postoperatively
Description: Using a Numeric Rating Scale, patients are asked to report their pain on a scale of 0 to 10 with 0 being no pain and 10 is the most imaginable. The variables will be presented as median and interquartile range.
Time Frame: 48 hours post surgical intervention
Measure: Median (Inter-Quartile Range); unit: scored on a scale
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 16 | 18
scored on a scale | 3 [0.25 to 3.75] | 2 [0.00 to 3.25]

3. Secondary Outcome: Quantitate the Amount of Opioid Medication Required to Provide Pain Relief-0 to 24 Hours Post Surgical Intervention
Description: To assess if either route (IV or ESP catheter) of lidocaine provided maximal pain relief when compared to its counterpart, the type and amount of medication provided the subject will be recorded. The opioid amounts required to provide relief during the first 24 hours will be tabulated in morphine equivalents. A comparison will be made between the two route to see if one route is optimal over the other. The variables will be presented as median and interquartile range.
Time Frame: First 24 hours post surgical intervention
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 30 | 30
Morphine Milligram Equivalents | 49.78 [29.52 to 72.57] | 39.00 [24.90 to 77.14]

4. Secondary Outcome: Quantitate the Amount of Opioid Medication Required to Provide Pain Relief-24 to 48 Hours Post Surgical Intervention
Description: To assess if either route (IV or ESP catheter) of lidocaine provided maximal pain relief when compared to its counterpart, the type and amount of medication provided the subject will be recorded. The opioid amounts required to provide relief 24 and 48 hours post surgical intervention will be tabulated in morphine equivalents. A comparison will be made between the two route to see if one route is optimal over the other. The variables will be presented as median and interquartile range.
Time Frame: From 24 to 48 hours post surgical intervention
Measure: Median (Inter-Quartile Range); unit: Morphine Milligram Equivalents
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 30 | 30
Morphine Milligram Equivalents | 24.5 [13.32 to 48.75] | 22.5 [7.50 to 37.70]

5. Secondary Outcome: Pain Score at 24 Hours Postoperatively
Description: as for outcome 2
Time Frame: 24 hours post surgical intervention
Measure: Median (Inter-Quartile Range); unit: Scored on a scale 0-10
Groups:
- Intravenous-Administration of Lidocaine: Subject will receive a bolus of lidocaine at 2 mg/kg ideal body weight. This is followed by lidocaine infusion via intravenous route at 2 mg/kg/hr for 48 hours after sham catheter placement.
  Intravenous Administration of Lidocaine Post Cardiac Surgery: Lidocaine will be administered via intravenously. Initial dose will be at 2 mg/kg ideal body weight followed by dosing at 2 mg/kg/hr for 48 hours
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 18 | 23
Scored on a scale 0-10 | 3.5 [3 to 6] | 5.0 [3 to 6]

6. Secondary Outcome: Quantify the Number of Subjects Who Had Lidocaine Plasma Levels Greater Than 5 Micrograms/Milliliter.
Description: All subjects will receive lidocaine via intravenous administration or through erector spinae plane block bilateral catheters. Arterial plasma levels monitoring the concentration of lidocaine will be checked at regular intervals. The number of subjects who reach levels above 5 micrograms/milliliter at the 24-hour timepoint will be reported.
Time Frame: 24 hours post intervention
Measure: Count of Participants; unit: Participants
Groups:
- Intravenous-Administration of Lidocaine: Subject will receive a bolus of lidocaine at 2 mg/kg ideal body weight. This is followed by lidocaine infusion via intravenous route at 2 mg/kg/hr for 48 hours .
  Intravenous Administration of Lidocaine Post Cardiac Surgery: Lidocaine will be administered via intravenously. Initial dose will be at 2 mg/kg ideal body weight followed by dosing at 2 mg/kg/hr for 48 hours
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
Number analyzed (Participants) | 28 | 27
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: First 72 hours after surgical procedure
Description: The definition is as described by clinicaltrials.gov
Arm/Group | Erector Spinae Plane Block-Administration of Lidocaine | Intravenous-Administration of Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
Ours is a single center trial. This likely should be investigated at multiple institutions with different surgical anesthesia groups for proper validation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04995497/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT04995497/ICF_001.pdf